CLINICAL TRIAL: NCT04352023
Title: Comparison of Analgesic Efficacy After Major Surgery in Pancreatobiliary Cancers: Intravenous Patient-controlled Analgesia Versus Patient-controlled Epidural Analgesia
Brief Title: Analgesic Efficacy After Pancreatobiliary Surgery: Intravenous Versus Patient-controlled Epidural
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Sang-Jae Park, Research Director, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCC-2017-0274
Record Dates: First submitted 2020-04-02; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Pancreatic Cancer; Biliary Tract Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms | interventions — Analgesia, Patient-Controlled

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial, prospective, single institute Experimental: A IV-PCA group IV-PCA drug: Fentanyl 3000 mcg and Oxycodone 100 mg were mixed Normal saline 200 ml Procedure/Surgery: Patient-controlled analgesia Intravenous patient-controlled analgesia Patient-controlled epidural analgesia
  Experimental: B PCEA group PCEA drug: Morphine 5 mg and Ropivacaine 750 mg were mixed Normal saline 400 ml loading of preadministered Morphine 1 mg and Ropivacaine 11.25 mg Procedure/Surgery: Patient-controlled analgesia Intravenous patient-controlled analgesia Patient-controlled epidural analgesia
Who Masked: Participant, Care Provider, Investigator
Masking Description: 2, 4, 6 block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (IV-PCA group) (Experimental): IV-PCA drug: Fentanyl 3000 mcg and Oxycodone 100 mg were mixed Normal saline 200 ml
  Interventions: Procedure: Patient-controlled analgesia
- B (PCEA group) (Experimental): PCEA drug: Morphine 5 mg and Ropivacaine 750 mg were mixed Normal saline 400 ml
  loading of preadministered Morphine 1 mg and Ropivacaine 11.25 mg
  Interventions: Procedure: Patient-controlled analgesia

INTERVENTIONS:
Procedure: Patient-controlled analgesia — Intravenous patient-controlled analgesia Patient-controlled epidural analgesia

SUMMARY:
Prospective, single institute based, open label, double arm, randomized controlled trial Hypothesis: Pain control after resection of hepatobiliary tumors in patients with PCEA is more effective than in patients with IV-PCA.

DETAILED DESCRIPTION:
Postoperative pain control is important in helping patients who underwent abdominal surgery to recover and to live a normal life. There is a method of administering painless injections to relieve postoperative pain. Currently, IV-PCA is mostly used. However, this method has a disadvantage in that the dosage of the opioid-based analgesic is increased, and thus side effects may be concerned. By administering analgesics through an epidural route approached through the thoracic vertebrae rather than intravenous injection, effective post-operative pain control and less side effects can be expected in lesser amounts. This study prospectively compared the pain control effects of IV-PCA and PCEA in patients undergoing resection of hepatobiliary tumors at the National Cancer Center, revealing that PCEA is more effective in alleviating pain after surgery. It has a purpose. In addition, the investigators will investigate and compare clinical outcomes (first fart, dietary progression, postoperative complications, etc.) of the two patient groups and investigate the side effects of PCEA and complications related to the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatobiliary malignancies
* Anticipating open surgery
* Written concent

Exclusion Criteria:

* History of previous upper abdominal open surgery
* Psychiatric problems
* Cognitive impairment
* Chronic pain

Elimination Criteria

* Rejected written concent
* Failure to follow instructions of doctor
* Stopped surgery due to peritoneal metastasis

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of analgesic efficacy after major surgery in pancreatobiliary cancers: Intravenous patient-controlled analgesia versus patient-controlled epidural analgesia | Day 2 postoperatively
  Comparison of pain scale (Numeric rating scale; minimum: 0, maximum: 10) of IV PCA and PCEA during ambulation on the day 2 postoperatively; Scale 0 means no pain and scale 10 means most painful

SECONDARY OUTCOMES:
Investigation and comparison of pain and clinical progress during rest after surgery, side effects of drugs administered to IV-PCA and PCEA, and complications related to PCEA procedure | 7 days
  Comparison of pain scale (Numeric rating scale; minimum: 0, maximum: 10) of IV PCA and PCEA during rest from the day 1 to 7 postoperatively; comparison of amount of totally infused analgesics, serum level of troponin I on the day 1 postoperatively, and incidence of postoperative complications between the two groups; investigation of PCEA-related complications and adverse effects of analgesics

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 3 years from the study completion date